CLINICAL TRIAL: NCT03796546
Title: A Prospective Trial to Investigate the Clinical Utility and Application of a Next Generation Sequencing Test for Pathogen Detection of Cerebral Spinal Fluid (CSF) Samples to Diagnose Pediatric Central Nervous System (CNS) Infections
Brief Title: Pediatric Infectious Disease Precision Medicine Using Sequencing Evaluation of CSF
Acronym: PIPSEC
Status: Completed | Type: Observational
Sponsor: IDbyDNA, Inc. (Industry)
Collaborators: Rady Children's Hospital, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: PIPSEC - 01
Record Dates: First submitted 2018-12-19; First posted 2019-01-08 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Infection; Meningitis
Keywords: Pediatric
MeSH Terms: conditions — Infections; Meningitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual cerebrospinal fluid collected for standard of care clinical diagnostic purposes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, multi-site, study to evaluate the diagnosis rate of DNA and RNA sequencing of cerebrospinal fluid for identification of pathogens directly in patients who have already had a spinal tap to evaluate for infection and were found to have a pleocytosis. Diagnostic rate and clinical utility of concurrent standard testing will be compared to diagnostic rate and clinical utility of DNA and RNA sequencing.

DETAILED DESCRIPTION:
IDbyDNA, Inc. has developed a robust sequencing reference database for viruses, bacteria, fungi and parasites and developed novel analysis methods to analyze next-generation (NGS) sequencing data to rapidly identify infectious agents. This technology suite, known as the Explify™ platform, holds the promise to improve patient care and efficiently guide provider treatment planning for those suffering from infectious disease.

The PIPSEC trial, developed by pediatric physicians specializing in genomic medicine, is intended to facilitate the acquisition of high quality and clinically annotated biospecimens for the purpose of research discovery. This project intends to advance metagenomics, microbial genetics, bioinformatics and data analytics, for pathogen detection utilizing cerebral spinal fluid (CSF) specimens to contribute to the diagnosis of infectious agents impacting the central nervous system among pediatric patients. Clinically annotated specimens will facilitate continued development and validation of the Explify test and its clinical utility for providers treating central nervous system (CNS) infections.

The primary objective is to assess clinical utility of the Explify test compared to concurrent standard of care testing to identify pathogens from CSF fluid within a pediatric patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-17 years of age (not yet 18)
* Clinical evaluation for CNS infection
* CSF white blood cell count (WBC) > 15 cells/µL when there are less than 5000 RBCs on same
* Admitted to a participating study site
* CSF obtained per standard protocol
* 1 mL of appropriately stored CSF is available following completion of all standard of care testing

Exclusion Criteria:

* CSF Red blood cell (RBC) count > 5000 cells/µL on same CSF sample as with pleocytosis
* Unable to obtain consent

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This project will enroll children who are having an evaluation for central nervous system (CNS) infection and have already had a lumbar puncture to obtain cerebrospinal fluid (CSF) to evaluate for infection and host immune response. As such enrolled patients will be undergoing an evaluation for suspected meningitis, encephalitis, ventriculitis and VP shunt infection.
  Patients in whom there is CSF remaining after standard testing has been obtained and who meet the other inclusion criteria will be approached for enrollment in the study.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic Rate | 24 months
  Comparison of the sensitivity, specificity, positive and negative predictive values of IDbyDNA NGS results with the Explify diagnostic platform compared with standard care.

SECONDARY OUTCOMES:
Clinical Utilization | 24 months
  Change of Management resulting from NGS diagnosis versus diagnosis based on standard of care. Change of Management is a binary (yes or no) based on assignments made by the PI or designee at each site using the following domains:
  * Diagnosis specific pharmacological treatment
  * Diagnosis specific management
  * Diagnosis specific supportive interventions A change in any of these domains will be considered a change of clinical management for utilization purposes.

OTHER OUTCOMES:
Post-Hoc Analysis - Economic Evaluation (1) | 24 months
  Economic evaluation of cost of standard of care testing compared to economic cost of NGS testing:
  Determination of what diagnosis made could have been made with best possible clinical tests currently available.
Post-Hoc Analysis - Economic Evaluation (2) | 24 months
  Cost analysis of what best available testing would have cost.
Post-Hoc Analysis - Host Response | 24 months
  RNA sequencing to determine if there is a specific host response to either specific infectious or noninfectious etiologies.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - CHOC Children's Hospital Orange County, Orange, California
  - Rady Children's Hospital, San Diego, California
  - Nicklaus Children's Hospital, Miami, Florida

IPD SHARING:
Plan to Share IPD: Undecided